CLINICAL TRIAL: NCT05446805
Title: The Impact of Depression and Preclinical Alzheimer Disease on Driving Among Older Adults (Depression and Driving)
Brief Title: Depression and Driving
Acronym: D&D
Status: Recruiting | Type: Observational
Sponsor: Ganesh Babulal (Other)
Responsible Party: Sponsor-Investigator, Ganesh Babulal, Associate Professor, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 202003209
Record Dates: First submitted 2022-06-03; First posted 2022-07-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Depression; Drive
MeSH Terms: conditions — Depression | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- depression: All participants will receive two one time PET scans with tracers AV1451 and PIB to detect tau and amyloid in the brain.
  Interventions: Drug: F 18 AV-1451 (Flortaucipir); Drug: [11C]-Pittsburgh Compound B ([11C]PiB)
- control: All participants will receive two one time PET scans with tracers AV1451 and PIB to detect tau and amyloid in the brain.
  Interventions: Drug: F 18 AV-1451 (Flortaucipir); Drug: [11C]-Pittsburgh Compound B ([11C]PiB)

INTERVENTIONS:
Drug: F 18 AV-1451 (Flortaucipir) — A dosage range between 6.5 - 10.0 mCi (240-370MBq) is planned for [18F] AV-1451. A PET-certified medical professional will prepare and administer the [18F] AV-1451tracer. Prior to the administration, the dosage will be assayed in a dose calibrator. The volume of 18F-AV-1451 dose should not be adjusted by adding normal saline to the syringe. Participants will receive a maximum intravenous bolus injection of 10.0 mCi of [18F] AV-1451 followed by a 10 mL flush of 0.9% sodium chloride (normal saline).
  Other Names: AV-1451
Drug: [11C]-Pittsburgh Compound B ([11C]PiB) — A dosage range between 6.0 - 20.0 mCi (222-740 MBq) is planned for [11C] PIB. A PET-certified medical professional will prepare and administer the [11C] PIB tracer. Prior to the administration, the dosage will be assayed in a dose calibrator and diluted with 0.9% sodium chloride (normal saline) up to a total 20 mL syringe volume. Participants will receive a maximum intravenous bolus injection of 20.0 mCi of [11C] PIB followed by a 10 mL 0.9% sodium chloride (normal saline) flush.
  Other Names: PIB

SUMMARY:
This project will assess how depression, preclinical AD, and antidepressants affect driving behavior in cognitively normal older adults (65 years).

DETAILED DESCRIPTION:
The long-term goal is to accurately identify who is at risk of decline in driving, to forecast when decline will occur, and to intervene before decline, thereby reducing the numbers of crashes, injuries, and death in older adults. The findings indicate that the long preclinical stage of Alzheimer disease (AD), as reflected in amyloid imaging and cerebrospinal fluid (CSF) biomarkers among cognitively normal participants, is associated with poorer driving performance on a standardized road test. This project will assess how depression, preclinical AD, and antidepressants affect driving behavior in cognitively normal older adults (65 years).

ELIGIBILITY:
Inclusion Criteria:

* Drive on average at least once per week
* Has a valid driver's license
* Willing to complete blood draw
* Willing to complete either lumbar puncture or PET imaging
* 65 years or older
* Speaks English

Exclusion Criteria:

* Not willing to complete blood draw and/or one other biomarker
* Less than 65 years of age
* Does not drive a vehicle/ is no longer actively driving

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: 70 participants will create a depressed cohort in which they must be determined to have active major depressive disorder (MDD) as defined by psychiatrist, Dr. Eric Lenze.
  70 participants will be cognitively normal (CDR 0) or cognitively abnormal (CDR 0.5 or 1) but will be considered control cohort.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Latitude via DRIVES chip | Daily for up to five years
  The latitude coordinate of the location of the vehicle being driven
Longitude via DRIVES chip | Daily for up to five years
  The Longitude coordinate of the location of the vehicle being driven
Vehicle Speed via DRIVES chip | Daily for up to five years
  The speed at which the vehicle being driven is moving.
Speed Limit via DRIVES chip | Daily for up to five years
  The posted speed limit for the location that participant is driving.
Difference via DRIVES chip | Daily for up to five years
  The difference between the speed at which the vehicle is moving and the posted speed limit for the location.
Event Name via DRIVES Chip | Daily for up to five years
  Name of the geofence in which participant had a driving event.
Address via DRIVES chip | Daily for up to five years
  Address of the location in which participant had a driving event.
Event Type via DRIVES chip | Daily for up to five years
  Enumeration describing the type of event: ignition on, heartbeat, ignition off, braking, acceleration, overspeeding, idling, low fuel, cornering, low battery event, diagnostic event triggered.
Event Time via DRIVES chip | Daily for up to five years
  Timestamp in GMT on which the event occurred.
Odometer Reading via DRIVES chip | Daily for up to five years
  Odometer reading of the vehicle.
Trip Distance via DRIVES chip | Daily for up to five years
  Total distance covered during the trip
Peak Speed via DRIVES chip | Daily for up to five years
  Highest speed attained by the vehicle during the trip.
Average Speed | Daily for up to five years
  Average trip speed of the vehicle.
Initial Speed via DRIVES chip | Daily for up to five years
  Speed at the beginning of the trip.
Final Speed via DRIVES chip. | Daily for up to five years
  Speed at the end of the trip.

SECONDARY OUTCOMES:
Trail Making A | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will test executive function.
Trail Making B | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will test executive function.
Montreal Cognitive Assessment (MoCA) Total | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will screen for cognitive impairment.
Category Fluency | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will test language ability.
Phonemic Fluency | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will test language ability.
Mini Mental Status Exam | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will screen for cognitive impairment.
Clinical Dementia Rating (CDR) Sum of Boxes | Annually for up to five years
  This will be tested annually in a private office setting using paper and pen assessments. This will test for cognitive impairment/dementia severity.

OTHER OUTCOMES:
Plasma based biomarker | Each participant will complete a blood draw within their first year of participation.
  Analyses of amyloid and tau burden among plasma samples
Cerebrospinal fluid biomarker | Each participant will complete an optional lumbar puncture within their first year of participation.
  Analyses of amyloid and tau burden among cerebrospinal fluid samples
Amyloid PET-based biomarker | Each participant will complete a PET scan with radiotracer PIB within their first year of participation.
  Amyloid measured by Pittburgh compound B
Tau PET-based biomarker | Each participant will complete a PET scan with radiotracer AV1451 within their first year of participation.
  Tau measured by AV1451

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Babulal, PhD, OTD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States